CLINICAL TRIAL: NCT05956639
Title: A Multi-center, Randomized, Open-label Clinical Trial Comparing a 6-month vs Long-term Course of Rezvilutamide With ADT Plus Chemotherapy in High Tumor Burden mHSPC
Brief Title: Comparing a 6-month vs Long-term Course of Rezvilutamide With ADT Plus Chemotherapy in mHSPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hua Lixin, M.D., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-258
Record Dates: First submitted 2023-06-20; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: Triple treatment regimen; mHPSC; Rezvilutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-month course of Rezvilutamide (Experimental): 6-month course of Rezvilutamide with ADT and chemotherapy
  Interventions: Drug: 6-month course of antiandrogen drugs
- Long-term course of Rezvilutamide (Active Comparator): Long-term course of Rezvilutamide with ADT and chemotherapy
  Interventions: Drug: Long-term course of antiandrogen drugs

INTERVENTIONS:
Drug: 6-month course of antiandrogen drugs — 6-month course of Rezvilutamide and ADT + chemotherapy
  Other Names: Rezvilutamide
  Arms: 6-month course of Rezvilutamide
Drug: Long-term course of antiandrogen drugs — Long-term course of Rezvilutamide and ADT + chemotherapy
  Other Names: Rezvilutamide
  Arms: Long-term course of Rezvilutamide

SUMMARY:
Primary Objective:

To explore whether a 6-month course of Rezvilutamide in the triple therapy regimen is non-inferior to long-term Rezvilutamide treatment in improving radiographic progression-free survival (rPFS) in patients with high tumor burden metastatic hormone-sensitive prostate cancer (mHSPC).

Secondary Objectives:

To evaluate and compare the time to prostate-specific antigen (PSA) progression, time to next bone-related event, time to initiation of subsequent anti-prostate cancer treatment, and objective response rate (ORR) between the 6-month and long-term course of Rezvilutamide with androgen deprivation therapy (ADT) plus docetaxel in patients with high tumor burden mHSPC.

To assess and compare the incidence of adverse events between the 6-month and long-term course of Rezvilutamide with ADT plus docetaxel in patients with high tumor burden mHSPC.

Exploratory Objectives:

To observe the circulating tumor cell status at 6 months, 12 months, 18 months, and 24 months in patients with high tumor burden mHSPC receiving the triple therapy regimen.

DETAILED DESCRIPTION:
Primary Study Endpoints:

Radiographic progression-free survival (rPFS)

Secondary Study Endpoints:

Time to prostate-specific antigen (PSA) progression Time to next bone-related event (including fractures, spinal cord compression, radiation therapy, or surgery targeting the bones) Time to initiation of subsequent anti-prostate cancer treatment Objective response rate (ORR) Quality of life assessment scores

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Age ≥ 18 years, male.
  2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
  3. Histologically or cytologically confirmed prostate adenocarcinoma without evidence of neuroendocrine or small cell features.
  4. High tumor burden, defined as having at least one of the following conditions: 1) Bone scan showing ≥4 bone metastatic lesions (with at least one site outside the pelvis or spine). 2) CT/MRI revealing visceral metastatic lesions (excluding lymph nodes).
  5. Planned to receive or maintain androgen deprivation therapy (ADT) during the study period, either by continuous LHRHa treatment or previous bilateral orchiectomy (surgical castration), concurrently with 6 cycles of docetaxel chemotherapy.
  6. Organ function levels must meet the following requirements:

     * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L.
     * Platelets (PLT) ≥ 100 × 10^9/L.
     * Hemoglobin (Hb) ≥ 90 g/L.
     * Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN).
     * Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
     * Aspartate aminotransferase (AST) ≤ 2.5 × ULN.
     * Blood urea nitrogen (BUN) (or urea) and creatinine (Cr) ≤ 1.5 × ULN.
     * Left ventricular ejection fraction (LVEF) ≥ 50%.
  7. Judged by the investigator to be able to comply with the trial protocol.
  8. Voluntarily participate in the clinical trial, understand the study procedures, and have signed the informed consent form.

Exclusion Criteria:

1. Prior treatment with ADT, chemotherapy, surgery, external beam radiation therapy, brachytherapy, radiopharmaceuticals, or investigational local therapies for prostate pain. However, the following cases are allowed for inclusion:

   * Up to 3 months of ADT (medical or surgical castration) with or without antiandrogen therapy prior to Cycle 1 Day 1 (C1D1) without evidence of radiographic disease progression (based on RECIST 1.1 criteria) or clinically significant PSA rise (defined as ≥50% increase from the lowest level after reaching castration levels of serum testosterone) before C1D1.
   * Transurethral prostatectomy or up to one course of palliative radiation therapy or surgery for symptomatic treatment of metastatic disease at least 4 weeks prior to C1D1. All adverse events related to these treatments must have improved to at least Grade 1 (according to NCI-CTCAE v4.03) before starting study treatment.
2. Prior use or planned use of second-generation androgen receptor antagonists (such as enzalutamide, apalutamide, darolutamide), abiraterone acetate, or other investigational drugs inhibiting testosterone synthesis for the treatment of prostate cancer during the study period.
3. Received the following treatments within 4 weeks before C1D1:

   * 5-alpha-reductase inhibitors (e.g., finasteride, dutasteride).
   * Estrogens, progestins, androgens, systemic corticosteroids (except for temporary use for allergic purposes).
   * Known herbal medicines with anti-prostate cancer or PSA-lowering effects (e.g., saw palmetto).
   * Participation in other clinical trials involving investigational treatments.
4. Confirmed brain tumor lesions on imaging.
5. Planned to receive any other anticancer treatment during the trial.
6. Known allergy or hypersensitivity to apalutamide, ADT, or chemotherapy components.
7. Presence of conditions that impede swallowing, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake and absorption.
8. History of seizures or occurrence of conditions that can induce seizures within 12 months before C1D1 (including transient ischemic attack, stroke, traumatic brain injury with altered consciousness requiring hospitalization).
9. Presence of active cardiac diseases within 6 months before C1D1, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and ventricular arrhythmias requiring medication.
10. Diagnosis of any other malignancy within 5 years before C1D1, except for completely resolved in situ cancer or malignancies with slow progression as determined by the investigator.
11. Active HBV or HCV infection (HBV viral load ≥ 10,000 copies/mL, HCV viral load ≥ 1,000 copies/mL).
12. History of immunodeficiency (including positive HIV test) or organ transplantation.
13. Unwillingness to use effective contraception during the entire study treatment period and for 30 days after the last dose.
14. Judged by the investigator to have conditions that pose a serious risk to patient safety, may confound study results, or may affect the patient's ability to complete the study (such as poorly controlled hypertension, severe diabetes, neurological or psychiatric diseases, etc.), or any other relevant circumstances.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
rPFS | 36 months
  Radiographic progression-free survival

SECONDARY OUTCOMES:
Time to prostate-specific antigen (PSA) progression | 36 months
  Time to PSA doubling on ADT + Rezvilutamide + Chemo
Time to next bone-related event | 36 months
  including fractures, spinal cord compression, radiation therapy, or surgery targeting the bones
Time to initiation of subsequent anti-prostate cancer treatment | through study completion, an average of 3 year
  Bone related treatment; Radiation therapy
Objective response rate (ORR) | 36 months
  PSA response, tumor burden shrink on radiographic reports
Quality of life assessment scores | 36 months
  Quality of life form with higher score indicating a better life experience under cancer condition

CONTACTS AND LOCATIONS:
Overall Officials: Lixxin Hua, Principal Investigator — Urology Dpt, First Affiliated Hospital of Nanjing Medical University
Locations (1):
- Urology dpt, First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05956639/Prot_000.pdf
  • Informed Consent Form (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05956639/ICF_001.pdf